CLINICAL TRIAL: NCT05672628
Title: The Feasibility, Usability, and Acceptability of Using the Oculus™ Virtual Reality Gaming Technology in Stroke Survivors for Upper Extremity and Cognitive Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: IoT and Aging in Place Joint Seed Grant (Unknown)
Responsible Party: Principal Investigator, Seema S Aggarwal, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SN-22-0838
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: rehabilitation; upper limb; stroke survivor
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Oculus VR (Experimental)
  Interventions: Device: Oculus VR

INTERVENTIONS:
Device: Oculus VR — During the first visit, the Oculus headset will be placed on the stroke survivor's head and demonstrate how to use the headset. participant will be then allowed to play a game using the hand controllers for up to 30 minutes. Finally, a copy of exercises for their home rehabilitation program will be provided. During the next rehabilitation visits, a trained research assistant will guide the stroke survivor with using the gaming headset. The session will be stopped every 20 minutes to make sure that the stroke survivor is feeling well and to give them a break. The stroke survivor may stop the session at any time. This session will last for an hour.

SUMMARY:
The purpose of this study is to test the (a) feasibility, (b) usability, and (c) acceptability of using the Oculus Virtual Reality (VR) for chronic stroke survivors who have mild-moderate cognitive and unilateral arm impairment to administer upper extremity and cognitive rehabilitation, to calculate the change in upper extremity and cognition scores on standardized measurements per standard of care and to qualitatively explore the impact of engaging caregivers in supporting the stroke survivor's rehabilitation and the impact of this engagement on the stroke survivor and caregiver dyad using semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke diagnosis within 6 months to 2 years of enrollment
* can read, write, comprehend, speak English
* willing and able to provide informed consent
* Caregivers must live in the home with the stroke survivor

Exclusion Criteria:

* do not have score ranges that indicate mild to moderate severity on the Montreal Cognitive Assessment (MoCA )(15-25) or other appropriate cognitive screening test selected by the speech language pathologist
* has aphasia, hemiopsia, and other neurological deficits that prevents the participant from being examined using MoCA or a modified MoCA, Fugl-Meyer Assessment - Upper Extremity (FM) (20-50)
* unstable while standing unassisted
* have a history of motion sickness/ vertigo/ dizziness/seizures, claustrophobia, blind/deaf, and cannot hold the controller in their affected arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema S Aggarwal, PhD, APRN, AGNP-C, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 individuals (16 dyads) were enrolled in total: 16 stroke survivor participants, each enrolled with a caregiver.
Period: Overall Study
Arm/Group | Oculus VR
Started | 32 (32 individuals (16 dyads) were enrolled in total: 16 stroke survivor participants, each enrolled with a caregiver.)
Completed | 32 (32 individuals (16 dyads) were enrolled in total: 16 stroke survivor participants, each enrolled with a caregiver.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oculus VR
Number analyzed (Participants) | 32
Age, Customized [Mean (Standard Deviation); unit: years] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads. Oculus VR arm = 16 dyads (16 stroke survivor participants + 16 caregivers= 32 participants).
  years
    Stroke Survivor Participant: number analyzed (Participants) | 16
    Stroke Survivor Participant | 50.31 (15.15)
    Caregiver: number analyzed (Participants) | 16
    Caregiver | 52.12 (10.81)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads. Oculus VR arm = 16 dyads (16 stroke survivor participants + 16 caregivers= 32 participants).
  Participants
    Stroke Survivor Participant: number analyzed (Participants) | 16
    Stroke Survivor Participant: Female | 5
    Stroke Survivor Participant: Male | 11
    Caregiver: number analyzed (Participants) | 16
    Caregiver: Female | 13
    Caregiver: Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads. Oculus VR arm = 16 dyads (16 stroke survivor participants + 16 caregivers= 32 participants).
  Participants
    Stroke Survivor Participant: number analyzed (Participants) | 16
    Stroke Survivor Participant: Black or African American | 8
    Stroke Survivor Participant: Hispanic/Latino | 2
    Stroke Survivor Participant: White | 6
    Caregiver: number analyzed (Participants) | 16
    Caregiver: Black or African American | 8
    Caregiver: Hispanic/Latino | 1
    Caregiver: White | 7
Region of Enrollment [Number; unit: participants]
  United States | 32
Level of Education [Count of Participants; unit: Participants] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads. Oculus VR arm = 16 dyads (16 stroke survivor participants + 16 caregivers= 32 participants).
  Participants
    Stroke Survivor Participant: number analyzed (Participants) | 16
    Stroke Survivor Participant: Associates | 1
    Stroke Survivor Participant: Bachelors | 3
    Stroke Survivor Participant: High School/GED | 3
    Stroke Survivor Participant: Masters | 2
    Stroke Survivor Participant: PhD | 1
    Stroke Survivor Participant: Some College | 6
    Caregiver: number analyzed (Participants) | 16
    Caregiver: Associates | 2
    Caregiver: Bachelors | 5
    Caregiver: High School/GED | 0
    Caregiver: Masters | 2
    Caregiver: PhD | 1
    Caregiver: Some College | 6
Stroke Type [Count of Participants; unit: Participants] — Population: Data for this outcome measure were only collected from the 16 stroke survivor participants
  Participants
    number analyzed (Participants) | 16
    Ischemic | 9
    Intracerebral hemorrhage | 6
    Subarachnoid hemorrhage | 1
Number of Participants with a right sided stroke [Count of Participants; unit: Participants] — Population: Data for this outcome measure were only collected from the 16 stroke survivor participants
  Participants
    number analyzed (Participants) | 16
    (all) | 10
Number of Participants with a history of previous stroke [Count of Participants; unit: Participants] — Population: Data for this outcome measure were only collected from the 16 stroke survivor participants
  Participants
    number analyzed (Participants) | 16
    (all) | 6
Type of Internet [Count of Participants; unit: Participants] — Population: Data for this outcome measure were only collected from the 16 stroke survivor participants
  Participants
    number analyzed (Participants) | 16
    Wi-fi | 13
    DSL | 3
Daily use of electronics [Count of Participants; unit: Participants] — Population: Data for this outcome measure were only collected from the 16 stroke survivor participants
  Participants
    number analyzed (Participants) | 16
    3-4 hours | 3
    4-8 hours | 7
    More than 8 hours | 6
Gaming Devices Used Previously [Count of Participants; unit: Participants] — Population: Data for this outcome measure were only collected from the 16 stroke survivor participants
  Participants
    Virtual Headset: number analyzed (Participants) | 16
    Virtual Headset | 9
    Game Console: number analyzed (Participants) | 16
    Game Console | 14
    Computer/Laptop: number analyzed (Participants) | 16
    Computer/Laptop | 9
    Smart Phone: number analyzed (Participants) | 16
    Smart Phone | 13
    Arcade: number analyzed (Participants) | 16
    Arcade | 11
Relationship of Stroke Survivor to Caregiver [Count of Participants; unit: Participants] — Relationship reflects how the stroke survivor is related to their enrolled caregiver. Population: Includes all 16 stroke survivor participants.
  Participants
    number analyzed (Participants) | 16
    Child of Caregiver | 1
    Friend of Caregiver | 1
    Parent of Caregiver | 3
    Sibling of Caregiver | 3
    Spouse of Caregiver | 8

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by the Number of Sessions Attended
Description: The minimum number of sessions expected for a user are 2 per week (8 sessions)
Time Frame: end of intervention( about 4 weeks from baseline)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
sessions | 11.06 (1.12)

2. Primary Outcome: Feasibility as Assessed by the Time Spent Using the Oculus VR
Description: the minimum time spent playing Job Simulator is 1 hour (60 minutes) per week. (240 minutes through the end of the study)
Time Frame: end of intervention( about 4 weeks from baseline)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
minutes | 785 (98.83)

3. Primary Outcome: Usability as Assessed by the Score on the System Usability Scale (SUS)
Description: The System Usability Scale (SUS) was used to assess the usability of the technology. Total score ranges from 10 to 50, with a higher score indicating greater usability.
Time Frame: end of intervention( about 4 weeks from baseline)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 32 (1.75)

4. Primary Outcome: Usability as Assessed by the Score on the Presence Questionnaire (PQ)
Description: The Presence Questionnaire (PQ), total score ranges from 29 to 87, with a higher score indicating greater usability.
Time Frame: end of intervention( about 4 weeks from baseline)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 75.86 (6.8)

5. Primary Outcome: Cognition as Assessed by the Montreal Cognitive Assessment (MoCA)
Description: Total score on the Montreal Cognitive Assessment (MoCA) range from 0 to 30, with a higher score indicating a better outcome.
Time Frame: Baseline
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 23.21 (4.88)

6. Primary Outcome: Cognition as Assessed by the Montreal Cognitive Assessment (MoCA)
Description: as for outcome 5
Time Frame: end of intervention (about 4 weeks from baseline)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 23.25 (3.59)

7. Primary Outcome: Limb Function as Assessed by the Action Research Arm Test (ARAT)
Description: Total score on the Action Research Arm Test (ARAT), ranging from 0 to 57, with higher scores indicating better upper limb function.
Time Frame: Baseline
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 19.37 (21.59)

8. Primary Outcome: Limb Function as Assessed by the Action Research Arm Test (ARAT)
Description: as for outcome 7
Time Frame: end of intervention( about 4 weeks from baseline)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 20.68 (21.13)

9. Primary Outcome: Arm Impairment as Assessed by Fugl Meyer - Upper Extremity Assessment
Description: Total score on the Fugl-Meyer Assessment - Upper Extremity (FMA-UE), ranges from 0 to 66, with higher scores indicating better arm function.
Time Frame: Baseline
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 30.56 (14.99)

10. Primary Outcome: Arm Impairment as Assessed by Fugl Meyer - Upper Extremity Assessment
Description: as for outcome 9
Time Frame: end of intervention( about 4 weeks from baseline)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 31.25 (19.26)

11. Primary Outcome: Burden of Caregivers in Supporting the Stroke Survivor as Assessed by the Burden Scale for Family Caregivers - Short Version
Description: Total score on the Burden Scale for Family Caregivers - short version, ranges from 0 to 30, with a higher score indicating more burden
Time Frame: Baseline
Population: Includes data for all 16 caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 13 (8.53)

12. Primary Outcome: Burden of Caregivers in Supporting the Stroke Survivor as Assessed by the Burden Scale for Family Caregivers - Short Version
Description: as for outcome 11
Time Frame: end of intervention( about 4 weeks from baseline)
Population: Includes data for 14 caregivers. Data were not collected for 2 caregivers because they did not fill out the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
score on a scale | 13.83 (7.55)

13. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: Total score on the Simulator Sickness Questionnaire (SSQ) questionnaire ranges from 16 to 64, a higher score indicating more cybersickness
Time Frame: Baseline
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 16.69 (1.35)

14. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 1 (week 1 day 1)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 16.38 (0.72)

15. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 2 (week 1 day 2)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 16.33 (0.72)

16. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 3 (week 1 day 3)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 16.25 (0.62)

17. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 4(week 2 day 1)
Population: Includes data for all 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 16.17 (0.72)

18. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 5 (week 2 day 2)
Population: Includes data for 15 stroke survivor participants. 1 participant did not attend the session therefore, data were not collected for 1 participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
score on a scale | 16.11 (0.33)

19. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 6 (week 2 day 3)
Population: Includes data for 14 stroke survivor participants. 2 participants did not attend the session therefore, data were not collected for 2 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
score on a scale | 16.33 (0.71)

20. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 7 (week 3 day 1)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
score on a scale | 16 (0)

21. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 8 (week 3 day 2)
Population: Includes data for 12 stroke survivor participants. 4 participants did not attend the session therefore, data were not collected for 4 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 12
score on a scale | 16.14 (0.38)

22. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 9 (week 3 day 3)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 12
score on a scale | 16.17 (0.41)

23. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 10 (week 4 day 1)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
score on a scale | 16.33 (0.58)

24. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 11 (week 4 day 2)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
score on a scale | 16.25 (0.5)

25. Primary Outcome: Acceptability (Ease of Use) as Assessed by the Score on the Simulator Sickness Questionnaire (SSQ) Questionnaire
Description: as for outcome 13
Time Frame: Session 12 (week 4 day 3)
Population: Includes data for 16 stroke survivor participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
score on a scale | 16 (0)

26. Secondary Outcome: Impact of the Rehabilitation on the Participant as Assessed by the Number of Themes Derived From the Qualitative Interview
Description: In-person, in-depth interviews will be conducted following completion of a virtual reality (VR) intervention using the Oculus Quest 2 headset for post-stroke rehabilitation. Interviews will be transcribed verbatim and a qualitative analytic process will be used to identify common themes. A codebook will be developed based on analysis of the transcripts. This outcome reflects the number of themes derived from the interviews.
Time Frame: Baseline
Population: Includes data from all 16 stroke survivor participants.
Measure: Number; unit: themes
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
themes | 5

27. Secondary Outcome: Impact of the Rehabilitation on the Caregiver as Assessed by Number of Themes Derived From the Qualitative Interview
Description: as for outcome 26
Time Frame: end of intervention( about 4 weeks from baseline)
Population: includes data for all 16 caregivers.
Measure: Number; unit: themes
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
themes | 5

28. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 1 (week 1 day 1)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 14

29. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 2 (week 1 day 2)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 8

30. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 3 (week 1 day 3)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 5

31. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 4(week 2 day 1)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 8

32. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 5 (week 2 day 2)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 5

33. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 6 (week 2 day 3)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
Participants | 6

34. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 7 (week 3 day 1)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 4

35. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 8 (week 3 day 2)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 12
Participants | 2

36. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 9 (week 3 day 3)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 12
Participants | 3

37. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 10 (week 4 day 1)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
Participants | 2

38. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 11 (week 4 day 2)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 2

39. Secondary Outcome: Number of Subjects Who Have Received Occupational Therapy
Time Frame: Session 12 (week 4 day3 )
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 1

40. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 1 (week 1 day 1)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 13

41. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 2 (week 1 day 2)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 7

42. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 3 (week 1 day 3)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 3

43. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 4(week 2 day 1)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 7

44. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 5 (week 2 day 2)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 3

45. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 6 (week 2 day 3)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
Participants | 6

46. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 7 (week 3 day 1)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 3

47. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 8 (week 3 day 2)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 12
Participants | 2

48. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 9 (week 3 day 3)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 12
Participants | 3

49. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 10 (week 4 day 1)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
Participants | 2

50. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 11 (week 4 day 2)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 2

51. Secondary Outcome: Number of Subjects Who Have Received Physical Therapy
Time Frame: Session 12 (week 4 day3 )
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 1

52. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 1 (week 1 day 1)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 11

53. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 2 (week 1 day 2)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 2

54. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 3 (week 1 day 3)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 2

55. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 4(week 2 day 1)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 3

56. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 5 (week 2 day2)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 1

57. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 6 (week 2 day 3)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
Participants | 2

58. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 7 (week 3 day 1)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 1

59. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 8 (week 3 day 2)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 12
Participants | 0

60. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 9 (week 3 day 3)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 12
Participants | 1

61. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 10 (week 4 day 1)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 14
Participants | 1

62. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 11 (week 4 day 2)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 15
Participants | 1

63. Secondary Outcome: Number of Subjects Who Have Received Speech Therapy
Time Frame: Session 12 (week 4 day 3)
Population: Includes data for all 16 stroke survivor participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oculus VR
Number analyzed (Participants) | 16
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: Adverse events were collected and reported only for the 16 stroke survivor participants. The 16 Caregiver participants did not undergo adverse event monitoring as they did not receive the intervention.
Arm/Group | Oculus VR
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 6/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oculus VR (N=16)
General Discomfort (General disorders) | 3 (11)
Fatigue (General disorders) | 2 (2)
Difficulty Focusing (Nervous system disorders) | 2 (2)
Increased Salivation (Gastrointestinal disorders) | 1 (2)
Difficulty Concentrating (Nervous system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT05672628/Prot_SAP_000.pdf